CLINICAL TRIAL: NCT00508001
Title: A Randomised, Double-blind, Parallel Group, Multi-centre, Phase II Study to Assess the Efficacy and Safety of Best Support Care (BSC) Plus ZD6474(Vandetanib) 300 mg, BSC Plus ZD6474(Vandetanib) 100 mg, and BSC Plus Placebo in Patients With Inoperable Hepatocellular Carcinoma (HCC)
Brief Title: Phase II Study of Best Support Care (BSC) Plus ZD6474(Vandetanib) in Patients With Inoperable Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4200C00072
Record Dates: First submitted 2007-07-25; First posted 2007-07-27 (Estimated); Results first posted 2012-07-17 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-08

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Hepatocellular carcinoma; Advanced solid, malignant tumour
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasms | interventions — vandetanib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): Best Supportive Care + Placebo
  Interventions: Drug: Best Supportive Care
- 2 (Experimental): Best Supportive Care + ZD6474 100 mg
  Interventions: Drug: Vandetanib
- 3 (Experimental): Best Supportive Care + ZD6474 300 mg
  Interventions: Drug: Vandetanib

INTERVENTIONS:
Drug: Vandetanib — ZD6474 300mg
  Other Names: Zactima; ZD6474
  Arms: 3
Drug: Vandetanib — ZD6474 100 mg
  Other Names: Zactima; ZD6474
  Arms: 2
Drug: Best Supportive Care — Placebo + Best Supportive Care
  Arms: 1

SUMMARY:
This is a multi-centre, phase II study to assess the efficacy and safety of ZD6474 in patients with Child-Pugh class A, inoperable HCC. This study comprises 2 phases, the primary treatment phase and the secondary treatment phase. The primary treatment phase is a randomised, double-blind, parallel-group phase II study to assess the efficacy and safety of ZD6474 300 mg plus best support care (BSC), ZD6474 100 mg plus BSC, and placebo plus BSC. The secondary treatment phase is an open-label expanded access program of ZD6474. In the primary treatment phase, patients will be randomised in a 1:1:1 ratio to receive ZD6474 300 mg plus BSC, ZD6474 100 mg plus BSC, or placebo plus BSC, respectively. Randomisation will be stratified on the basis of Cancer of the Liver Italian Programme (CLIP) tumour staging (CLIP score 0-2 versus 3-4). The primary treatment will continue until objective disease progression, according to Response Evaluation Criteria in Solid Tumours (RECIST) criteria, or until patients meet any other withdrawal or discontinuation criteria.The primary endpoint is tumour stabilisation rate, and the secondary endpoints are objective response rate, progression-free survival, and overall survival. The purpose of the secondary treatment phase is to expand the access of ZD6474 so that every patient who is enrolled into this study can have the chance to receive the active medicine.Once an individual patient has progressive disease in the primary treatment phase, the blind will be broken for this patient. If this patient is in the ZD6474 100 mg arm or placebo arm, the patient will be offered the secondary treatment with ZD6474 300 mg per day. If this patient is randomised to the ZD6474 300 mg arm, the study medication will be discontinued unless the patient wishes to remain the treatment, and the patient is to be followed up for survival.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and provide informed consent
* Histologically diagnosed HCC, OR clinically diagnosed HCC for patients with difficulty in obtaining histological diagnosis. A clinically diagnosed HCC should fulfil ALL the criteria below.

  * Chronic hepatitis B or C and/or evidence of liver cirrhosis
  * Presence of hepatic tumour(s) with image findings (sonography, CT scan, or MRI scan) compatible with HCC, and no evidence of other gastrointestinal tumours
  * A persistent elevation of serum a-fetoprotein level >= 400 ng/ml without any evidence of an existing a-fetoprotein-secreting germ cell tumour
* Locally advanced (for example, portal vein invasion, multiple nodules, or nodules in both lobes) or metastatic HCC with at least one measurable lesion by RECIST criteria that meets ANY the criteria below:

  * HCC not suitable to receive local therapy, including surgical resection, percutaneous ethanol injection (PEI), or transarterial chemo-embolization (TACE)
  * Disease recurred or was refractory to previous local therapy
  * Patients refused local therapy
* At least one measurable lesion by RECIST criteria. Tumour lesions treated previously with local radiotherapy, percutaneous ethanol injection, radiofrequency ablation, or transarterial embolization are NOT considered measurable.
* If they completed percutaneous ethanol injection, radiofrequency ablation, transarterial embolization, or cryotherapy at least 4 weeks prior to enrollment, patients must have subsequent progression or recurrence with at least one new measurable lesion that has not been treated with any local procedure.
* Karnofsky performance status >= 70
* Life expectancy >= 2 months
* Child-Pugh class A liver function
* Adequate bone marrow reserve, defined as white blood cell count >= 3,000/ml, and platelet count >= 75,000/ml
* Liver transaminases (AST and ALT) <= 5 times upper normal limits (UNLs); serum bilirubin <= 1.5 times UNL <= 2 mg/dL
* Serum creatinine <= 1.5 times UNL
* Negative pregnancy test for women of childbearing potential. Patients of childbearing age as well as his/her partner must use effective contraception during the study period unless they are surgically sterile or one year post-menopausal

Exclusion Criteria:

* Receiving concurrent anti-cancer therapy for HCC, which includes local therapy, chemotherapy, or other experimental therapy
* Prior systemic cytotoxic chemotherapy
* Prior transarterial chemo-embolization (TACE) or hepatic arterial infusion (HAI), with any of the following conditions for those patients who have any target lesions in the liver:

  * More than 5 TACE or HAI sessions undergone prior to enrollment
  * The cumulative doses of doxorubicin > 120 mg/m2, mitomycin-C > 24 mg/m2, cisplatin > 120 mg/m2, or 5-fluorouracil > 2400 mg/m2
  * Details of the TACE or HAI regimens are not available in the chart
* (Note: The number of sessions of prior TACE or HAI will not be limited for patients who have no target lesion in the liver).
* Local treatment including radiotherapy (except palliative radiotherapy), percutaneous ethanol injection, radiofrequency ablation, transarterial embolization, or cryotherapy completed within 4 weeks prior to enrollment
* Prior therapy targeting VEGF or EGF signalling pathways, including but not limited to bevacizumab, cetuximab, gefitinib, erlotinib, or sorafenib.
* Prior thalidomide therapy is not allowed but for patients who stop thalidomide due to intolerability and meet either one of following condition can be included:

  * Patients who took thalidomide for no more than <= 3 days before enrolment
  * Patients who took thalidomide for > 3 days but <= 14 days and are confirmed clinically not responding to thalidomide. 14 days washout period is needed before enrolment.
* Laboratory results:

  * Serum potassium less than 4.0 mmol/L despite supplementation
  * Serum calcium (ionized or adjusted for albumin) or magnesium out of their normal ranges despite supplementation
* Esophagogastroduodenoscopy reveals lesions that are considered high risk of gastrointestinal bleeding
* Brain or leptomeningeal metastases
* History of HCC tumour rupture
* History of upper gastrointestinal bleeding within 1 year
* Current or recent (within 10 days prior to enrollment) users of full-dose oral or parenteral anti-coagulants
* Surgical procedures, open biopsy, or significant traumatic injury within 28 days prior to enrollment. Fine-needle aspiration, core biopsy, and central venous line placement must be done at least 7 days prior to enrollment. Incompletely healed surgical incision prior to enrollment.
* Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the investigator's opinion makes it undesirable for the patient to participate in the study or which would jeopardize compliance with the protocol.
* Clinically significant cardiac event such as myocardial infarction; New York Heart Association classification of heart disease > 2 within 3 months before entry; or other cardiac disease that, in the opinion of the investigator, increases the risk of ventricular arrhythmia.
* History of arrhythmia (multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia, or uncontrolled atrial fibrillation), which is symptomatic, requires treatment (CTCAE grade 3), or asymptomatic sustained ventricular tachycardia. Atrial fibrillation, if controlled on medication, will not be excluded.
* Previous history of QTc prolongation as a result of therapy with other medication that required discontinuation of that medication.
* Congenital long QT syndrome, or first-degree relative with unexplained sudden death under 40 years of age
* Presence of left bundle branch block
* QTc with Bazett's correction that is unmeasurable, or >= 480 msec on screening ECG
* Use of any concomitant medication that are generally accepted by authorities to have a risk of causing Torsades de Pointes within 2 weeks before enrollment (use of the concomitant medication that may be associated with Torsades de Pointes but lack substantial evidence of causing Torsades de Pointes is allowed, but the screening QTc must be less then 460 msec, and an additional ECG is required within the first 24 hours after the first dose of study medication is required).
* Use of any concomitant medication that induce CYP3A4 activity within 2 weeks before enrollment
* Use of interferon within 3 months before enrollment
* Hypertension not well controlled by medical therapy (systolic blood pressure greater than 160 mmHg or diastolic blood pressure greater than 100 mmHg)
* Currently active diarrhea that may affect the ability of the patient to absorb the ZD6474 or diarrhea due to intolerability
* Current pregnancy or breast-feeding
* Other previous or current malignancies within the last 5 years, with the exception of adequately treated cervical carcinoma in situ and basal cell or squamous cell carcinoma of the skin
* Receipt of any investigational agents within 30 days prior to commencing protocol treatment
* Any unresolved toxicity greater than CTC grade 2 from previous anti-cancer therapy
* Known hypersensitivity to ZD6474 or any of its excipients

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2007-07; Primary Completion 2008-11 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director Clinical Sciences & Operations, Study Director — Sanofi
Locations (3):
- Taiwan (3):
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 78 patients were recruited at medical clinic
Pre-assignment Details: 11 patients were screening failure due to inclusion criteria or exclusion criteria is not fulfilled
Groups:
- ZD6474 300: ZD6474 (Vandetanib) 300 mg ( one tablet per day, orally). plus Best Support Care
- ZD6474 100: ZD6474 (Vandetanib) 100 mg (one tablet per day, orally). plus Best Support Care
- Placebo: Placebo plus Best Support Care
Period: Overall Study
Arm/Group | ZD6474 300 | ZD6474 100 | Placebo
Started | 19 | 25 | 23
Secondary Treatment Phase | 0 | 13 | 16
Completed | 0 | 13 | 16
Not Completed | 19 | 12 | 7
Not completed — Adverse Event | 2 | 0 | 4
Not completed — condition under investigation worsened | 13 | 7 | 1
Not completed — Death | 0 | 1 | 1
Not completed — Withdrawal by Subject | 4 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ZD6474 300 | ZD6474 100 | Placebo | Total
Number analyzed (Participants) | 19 | 25 | 23 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (13.48) | 61.2 (13.36) | 57.3 (12.62) | 58.37 (13.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 20 | 55
  Male | 1 | 8 | 3 | 12
Child-Pugh Score [Number; unit: Participants] — Child-Pugh Scale is used to assess the prognosis of chronic liver disease. The total score employs five clinical measures of liver disease: severity of ascites and of encephalopathy, abnormality in the serum bilirubin, serum albumin and clotting times. Each measure is scored 1-3, with 3 indicating most severe derangement.
  The Total score ranges between 5 min to 15 max where lower score = less liver disease and higher score = chronic liver disease.
  The number of patients with Child-PughTotal score of 5 and 6 is presented.
  Participants
    Child-Pugh of 5 | 13 | 19 | 17 | 49
    Child-Pugh of 6 | 6 | 6 | 6 | 18
CLIP Score [Number; unit: Participants] — Cancer of the Liver Italian Programme (CLIP) is used to evaluate both tumour extension and remnant liver function with a score of min 0 to max 4. The CLIP score consists of 4 variables: Child-Pugh stage, tumour morphology, alpa-fetoprotein (AFP), and portal vein thrombosis. The higher the CLIP score the worse the survival.
  The number of patients with CLIP Total score of 0, 1, 2, 3 and 4 is presented.
  Participants
    CLIP 0 | 2 | 1 | 0 | 3
    CLIP 1 | 5 | 5 | 3 | 13
    CLIP 2 | 2 | 5 | 8 | 15
    CLIP 3 | 4 | 8 | 6 | 18
    CLIP 4 | 6 | 6 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Tumour Stabilisation Rate
Description: Tumour stabilisation rate calculated as percentage of patients with best objective tumour response (Complete Response, Partial Response or Stable Disease) for >=16 weeks based on Response Evaluation Criteria in Solid Tumours (RECIST).
  Complete Response - Disappearance of all target lesions; Partial Response - >=30% decrease in the sum of longest diameter of target lesions; Progressive Disease - >=20% increase in the sum of longest diameter of target lesions; Stable Disease - neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: After 16 weeks of treatment.
Population: The analysis has been performed in the Intent-To-Treat (ITT) population.
Measure: Number; unit: percentage of patients
Arm/Group | ZD6474 300 | ZD6474 100 | Placebo
Number analyzed (Participants) | 19 | 25 | 23
percentage of patients | 5.3 | 16.0 | 8.7

2. Secondary Outcome: Objective Response Rate
Description: Objective Response rate defined as percentage of patients with Complete Response [CR] or Partial Response [PR] based on Response Evaluation Criteria in Solid Tumours (RECIST).
  Partial response (PR) must have ≥ 30% decrease in the sum of longest diameter of all target lesions as assessed by Magnetic Resonance Imaging (MRI). Complete response (CR) must have disappearance of all target and non-target lesions as assessed by MRI.
Time Frame: After 16 weeks of treatment.
Population: The analysis has been performed in the Intent-To-Treat (ITT) population.
Measure: Number; unit: percentage of patients
Arm/Group | ZD6474 300 | ZD6474 100 | Placebo
Number analyzed (Participants) | 19 | 25 | 23
percentage of patients | 0 | 0 | 0

3. Secondary Outcome: Progression-free Survival
Description: Progression-free survival defined as the period from date of randomization(start of treatment) to date of disease progression or death.
Time Frame: from the date of randomisation to the date of documented disease progression or death for any cause
Population: The analysis has been performed in the Intent-To-Treat (ITT) population.
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | ZD6474 300 | ZD6474 100 | Placebo
Number analyzed (Participants) | 19 | 25 | 23
Days | 32 (29) [29 to 108] | 53 (29) [29 to 57] | 29 (28) [28 to 57]

4. Secondary Outcome: Overall Survival
Description: Overall survival defined as the time from randomization (start of treatment) until death from any cause.
Time Frame: assessed up to 360 days
Population: The analysis performed in the intent-To-Treat population.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | ZD6474 300 | ZD6474 100 | Placebo
Number analyzed (Participants) | 19 | 25 | 23
Days | 181 [117 to 290] | 175 [137 to 309] | 130 [93 to 180]

ADVERSE EVENTS:
Arm/Group | ZD6474 300 | ZD6474 100 | Placebo
Serious Adverse Events (participants affected / at risk) | 6/19 | 4/25 | 4/23
Other Adverse Events (participants affected / at risk) | 18/19 | 24/25 | 21/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ZD6474 300 (N=19) | ZD6474 100 (N=25) | Placebo (N=23)
Myocardial Ischaemia (Cardiac disorders) | 1 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal Varices Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Mucosal Inflammation (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Hepatic Failure (Hepatobiliary disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Weight Decreased (Injury, poisoning and procedural complications) | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 0 | 0 | 1
Stevens-Johnson Syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ZD6474 300 (N=19) | ZD6474 100 (N=25) | Placebo (N=23)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2
Deficiency Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0
Vision Blurred (Eye disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 9 | 7
Constipation (Gastrointestinal disorders) | 2 | 3 | 5
Vomiting (Gastrointestinal disorders) | 2 | 3 | 5
Nausea (Gastrointestinal disorders) | 0 | 3 | 3
Abdominal Distension (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 2
Gastric Ulcer (Gastrointestinal disorders) | 2 | 0 | 0
Mouth Ulceration (Gastrointestinal disorders) | 2 | 0 | 0
Periodontitis (Gastrointestinal disorders) | 0 | 2 | 0
Anal Fissure (Gastrointestinal disorders) | 1 | 0 | 0
Dry Mouth (Gastrointestinal disorders) | 1 | 1 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0 | 0
Frequent Bowel Movements (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal Disorder (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Irritable Bowel Syndrome (Gastrointestinal disorders) | 1 | 0 | 1
Lip Ulceration (Gastrointestinal disorders) | 1 | 0 | 0
Oral Pain (Gastrointestinal disorders) | 1 | 0 | 0
Peptic Ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Rectal Tenesmus (Gastrointestinal disorders) | 1 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 0
Fatigue (General disorders) | 1 | 3 | 1
Oedema Peripheral (General disorders) | 1 | 1 | 3
Pyrexia (General disorders) | 2 | 4 | 3
Mucosal Inflammation (General disorders) | 1 | 3 | 0
Malaise (General disorders) | 1 | 1 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 4 | 2
Bronchitis (Infections and infestations) | 1 | 2 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0
Post Procedural Complication (Injury, poisoning and procedural complications) | 0 | 0 | 2
Limb Injury (Injury, poisoning and procedural complications) | 1 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 1
Electrocardiogram Qt Prolonged (Injury, poisoning and procedural complications) | 2 | 2 | 1
Weight Decreased (Injury, poisoning and procedural complications) | 1 | 1 | 3
Aspartate Aminotransferase Increased (Injury, poisoning and procedural complications) | 1 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 4 | 3 | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 5
Headache (Nervous system disorders) | 1 | 0 | 0
Poor Quality Sleep (Nervous system disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 4 | 5
Anxiety (Psychiatric disorders) | 1 | 0 | 2
Nocturia (Renal and urinary disorders) | 0 | 0 | 3
Dysuria (Renal and urinary disorders) | 1 | 1 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0
Scrotal Ulcer (Reproductive system and breast disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 3
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 9 | 6 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 5 | 2
Acne (Skin and subcutaneous tissue disorders) | 4 | 4 | 4
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 1 | 3 | 0
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Rash Erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash Macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin Plaque (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 2 | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.